CLINICAL TRIAL: NCT06725433
Title: NiDor-study: a Randomized Controlled Trial Comparing Nissen and Dor Fundoplication in Hiatal Hernia Repair
Brief Title: Nissen Versus Dor Hiatal Hernia Repair
Acronym: NiDor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUH5204535
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Hiatal Hernia; Paraesophageal Hernia; Recurrence
MeSH Terms: conditions — Hernia, Hiatal; Recurrence | interventions — Fundoplication

STUDY DESIGN:
Intervention Model Description: Prospective open label randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nissen fundoplication (Active Comparator): Hiatal hernia repair and Nissen (posterior 360-degree) fundoplication
  Interventions: Procedure: Nissen fundoplication
- Dor fundoplication (Experimental): Hiatal hernia repair and Dor (anterior 180-degree) fundoplication
  Interventions: Procedure: Dor fundoplication

INTERVENTIONS:
Procedure: Nissen fundoplication — Hiatal hernia repair and Nissen fundoplication
  Arms: Nissen fundoplication
Procedure: Dor fundoplication — Hiatal hernia repair and Dor fundoplication
  Arms: Dor fundoplication

SUMMARY:
Hiatal hernia can present with a wide range of symptoms. An usual surgical repair technique usually includes Nissen fundoplication, while other procedures are less frequently employed. However, recurrence and reoperation rates remain high. This randomized controlled trial aims to compare the efficacy of Nissen and Dor fundoplication in preventing hiatal hernia recurrence and reducing the risk of reoperation

Participants undergoing minimally invasive hiatal hernia repair will be randomly assigned to either Nissen or Dor fundoplication. Postoperatively at 12 months, anatomical recurrence rates based on computed tomography scans and symptomatic recurrence rates, anti-reflux medication use, GERD-related quality of life, and dysphagia symptoms will be assessed. A subsequent long-term follow-up study will conducted afterwards utilizing national registry data to evaluate reoperation rates and anti-reflux medication use

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Type II-IV hiatal hernia, confirmed by radiology or endoscopy
* Scheduled for mini-invasive hiatal hernia repair
* Emergency mini-invasive surgery for hiatal hernia
* The informed consent is acquired

Exclusion Criteria:

* Recurrent hiatal hernia
* Need for esophageal lengthening procedure (Collis)
* Gangrene or need for any resection during (emergency) surgery
* Need for laparotomy or thoracotomy/thoracoscopy
* No written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Anatomical recurrence of hiatal hernia | 12 months after the surgery
  Computed tomography based recurrence after Nissen versus Dor fundoplication
Symptomatic recurrence of hiatal hernia | 12 months after the surgery
  Anatomical recurrence with questionnaire based gastroesophageal reflux disease (GERD) or dysphagia symptoms, or need for reoperation for recurrence

SECONDARY OUTCOMES:
Symptomatic versus asymptomatic recurrence rates | 12 months
  Symptomatic versus asymptomatic recurrence rates at 12 months
Reoperation rates | 20 years
  Reoperation rates at 3-, 5-, 10- and 20-years following the surgery
Managing GERD symptoms with Nissen vs Dor fundoplication | 12 months
  The efficacy of Nissen vs Dor fundoplication techniques in improving the Gastroesophageal Reflux Disease-Health Related Quality of Life instrument (GERD-HRQL) scores at 12 months. Minimum score 0 = no symptoms, maximum score 75 = worst symptoms.
Dysphagia symptoms after Nissen vs Dor fundoplication | 12 months
  The effect of different fundoplication techniques on dysphagia symptoms assessed by Eating Assessment Tool (EAT-10 ) at 12 months. Score range from 0 to 40 with higher scores indicating more severe dysphagia.
Hiatal hernia size and recurrence rates | 12 months
  The association between hiatal hernia size and recurrence rates. During surgery, the left-to-right and posterior-to-anterior dimensions of the hiatal opening, as well as whether more than 30% of stomach is herniated , will be recorded. These measurements will then be compared to postoperative recurrence rates."
Proton pump inhibitor usage | 20 years
  Proton pump inhibitor usage will be assessed at 1- 3-, 5-, 10- and 20-years after surgery
The impact of Body Mass Index on recurrence and reoperation rates | 20 years
  The impact of initial Body Mass Index (BMI, kg/m^2) on the recurrence rates (12 months) and reoperation rates (1-, 3-, 5-, 10- and 20-years)
The impact of age on recurrence and reoperation rates | 20 years
  The impact of subject age (years) on the recurrence rates (12 months) and reoperation rates (1-, 3-, 5-, 10- and 20-years)
The impact of albumin level on recurrence and reoperation rates | 20 years
  The impact of albumin level (g/l) on the recurrence rates (12 months) and reoperation rates (1-, 3-, 5-, 10- and 20-years)

CONTACTS AND LOCATIONS:
Overall Officials: Ville Palomäki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No